CLINICAL TRIAL: NCT03774784
Title: A Study of the Natural History of Leukocyte Chemotactic Factor 2 Amyloidosis (ALECT2) Disease
Status: Terminated | Type: Observational
Why Stopped: The study was terminated due to the impacts of COVID-19 on patient safety and enrollment.
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-LECT2-NT-001
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Amyloidosis; Leukocyte Chemotactic Factor 2 Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALECT2 Disease

SUMMARY:
The purpose of this study is to characterize the natural history of leukocyte chemotactic factor 2 amyloidotic (ALECT2) disease. In this observational study participants with ALECT2 disease will be enrolled. Participants, who have already reached end-stage renal disease (ESRD), will provide retrospective chart review data and biological specimens at baseline only. Other participants, in addition to retrospective chart review, will be followed prospectively.

DETAILED DESCRIPTION:
Refer to www.studyALECT2.com

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 years or older;
* Renal biopsy-proven diagnosis of ALECT2;
* For patients with kidney disease that could be due to ALECT2, a renal biopsy may be obtained to confirm ALECT2 diagnosis.

Exclusion Criteria:

- There are no exclusion criteria for this observational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with biopsy-proven ALECT2.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) from Baseline Up to End of Study (Month 48) | Baseline (Day 1), Months 6, 12, 18, 24, 30, 36, 42 and 48
Time to End-Stage Renal Disease (ESRD) | From baseline to end of study (Month 48)

SECONDARY OUTCOMES:
Level of Leukocyte Chemotactic Factor 2 (LECT2) Messenger Ribonucleic Acid (mRNA) in Blood | Baseline (Day 1), Months 6, 12, 18, 24, 30, 36, 42 and 48
Level of LECT2 mRNA in Urine | Baseline (Day 1), Months 12, 24, 36 and 48
Level of LECT2 Protein in Blood | Baseline (Day 1), Months 6, 12, 18, 24, 30, 36, 42 and 48
Level of LECT2 Protein in Urine | Baseline (Day 1), Months 12, 24, 36 and 48
Percentage of Participants With Proteinuria | Baseline (Day 1), Months 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Friedman, MD, Study Director — Alnylam Pharmaceuticals
Locations (30):
- United States (15):
  - Clinical Trial Site, Scottsdale, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Indianapolis, Indiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Albuquerque, New Mexico
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, St. George, Utah
- Egypt (4):
  - Clinical Trial Site, Al Mansurah
  - Clinical Trial Site, Alexandria
  - Clinical Trial Site, Asyut
  - Clinical Trial Site, Cairo
- India (5):
  - Clinical Trial Site, Chandigarh
  - Clinical Trial Site, Ludhiāna
  - Clinical Trial Site, Manipal
  - Clinical Trial Site, Nadiād
  - Clinical Trial Site, Tamil Nadu
- Clinical Trial Site, Kuala Lumpur, Malaysia
- Mexico (4):
  - Clinical Trial Site, Mexicali, Baja
  - Clinical Trial Site, México, Mexico DF
  - Clinical Trial Site, Culiacán, Sinaloa
  - Clinical Trial Site, Monterrey
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No